CLINICAL TRIAL: NCT02071381
Title: A Randomized, Open Label, Single-Dose, 6-sequence, 3-period, Crossover Study to Evaluate a Pharmacokinetic Drug Interaction Between DW330SR and DW1030 in Healthy Male Subjects
Brief Title: Phase 1 Study of DDI Between DW330SR and DW1030 in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daewon Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: DW340-1001
Record Dates: First submitted 2014-02-21; First posted 2014-02-25 (Estimated); Last update posted 2015-03-30 (Estimated); Status verified 2014-01

CONDITIONS: Healthy

ARMS (3):
- A (Experimental): only DW330SR 45mg
  Interventions: Drug: DW330SR 45mg
- B (Experimental): only DW1030 75mg
  Interventions: Drug: DW1030 75mg
- C (Experimental): DW330SR 45mg and DW1030 75mg
  Interventions: Drug: DW330SR 45mg; Drug: DW1030 75mg

INTERVENTIONS:
Drug: DW330SR 45mg
  Arms: A; C
Drug: DW1030 75mg
  Arms: B; C

SUMMARY:
The purpose of this study is to evaluate drugs interactions to compare pharmacokinetics in groups of monotherapy DW330SR, monotherapy DW1030, and coadministration DW330SR and DW1030

ELIGIBILITY:
Inclusion Criteria:

* Healthy Adult males aged 20~40 years at screening visit
* Subjects with range of 19 kg/m2 ~ 27 kg/m2 as BMI measurements at screening visit
* Subjects with BP range of below:

  90 mmHg ≤ Systolic BP ≤ 140 mmHg 50 mmHg ≤ Diastolic BP ≤ 90mmHg
* Subjects who voluntarily agreed with written consent that be able to understand the objective, method of the study, the characteristics of investigational drug, and comply with the reguirement of the study

Exclusion Criteria:

* Subjects with clinically significant disease or history such as Liver, kidney, gastrointestinal, respiratory, musculoskeletal, endocrine, nervous psychiatric, blood tumor system and cardiovascular. (In particular, bronchial asthma, severe hepatic, renal failure, severe blood disorders, severe myasthenia gravis, cardiac dysfunction, peptic ulcer, etc.)
* Subjects with history of gastrointestinal disease (ex, Chrones dz, peptic ulcer, etc) affect the absorption of Investigational drugs or history of surgery (except for a simple appendectomy or hernia surgery)
* Subjects with hypersensitivity reaction or clinically significant disease in drugs (Aspirin, NSAID and antibiotics) including ingredient of DW330SR and DW1030 and Food

Ages: 20 Years to 40 Years | Sex: Male
Age Groups: Adult
Dates: Start 2014-04; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Trans-OH as Main Metabolites of DW330SR, DW330SR, Cmax, AUClast of DW1030 | -28 ~ -2day(screening), -1day, 1day, 2day

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center IRB, Seoul, South Korea